CLINICAL TRIAL: NCT07122414
Title: A Phase I/II, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-Tumor Activity of Intravesical FL115 Alone or in Combination With BCG in Subjects With Non-Muscle Invasive Bladder Cancer, Including Dose Escalation and Cohort Expansion
Brief Title: A Study of Intravesical FL115 Alone or in Combination With BCG in Non-Muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Forlong Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL115-103
Record Dates: First submitted 2025-07-21; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FL115 and BCG (Experimental)
  Interventions: Drug: FL115; Drug: FL115+BCG

INTERVENTIONS:
Drug: FL115 — FL115 single agent dose escalation,
Drug: FL115+BCG — FL115 in combination with BCG

SUMMARY:
The study is to evaluate the safety and tolerability of intravesical FL115 alone or in combination with BCG in the patients with NMIBC, and to determine the RP2D of FL115 in combination with BCG.

To evaluate the preliminary efficacy of FL115 alone or in combination with BCG in the treatment of NMIBC.

The study consists of three parts: FL115 monotherapy dose escalation (Phase Ia), FL115 combined with BCG dose escalation (Phase Ib), and FL115 combined with BCG cohort expansion (Phase II).

Each subject will receive FL115 alone or in combination with intravesical BCG, administered over three treatment periods: induction, enhanced induction/maintenance 1, and maintenance 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older.
2. Histologic confirmation of non-muscle invasive bladder cancer of the transitional cell carcinoma high-grade subtype (mixed histology tumors allowed if transitional cell histology is predominant histology).
3. Histologically confirmed presence of BCG-unresponsive CIS (with or without Ta or T1 disease) or histologically confirmed presence of BCG-unresponsive high-grade Ta or T1 disease.
4. Absence of resectable disease after transurethral resection (TURBT) procedures (residual carcinoma in situ (CIS) acceptable; patients with T1 tumors must undergo repeat resection and biopsy [inclusive of muscularis propria] if initial biopsy did not include muscularis propria). Patients with high-grade Ta and/or T1 disease should have complete resection before study treatment.
5. Subjects refuse or are judged by the investigator not suitable for radical cystectomy.
6. ECOG score 0-2.
7. Expected survival ≥ 2 years (judged by the investigator).
8. Adequate organ function.
9. Voluntary written informed consent and agree to comply with all protocol-specified procedures and follow-up evaluations.

Exclusion Criteria:

1.Prior Anti-Cancer Treatment History:

1. Have previously received IL-2 or IL-15 agonist therapy, including but not limited to rhIL-15 (NCI), ALT-803 (FL-115), and NKTR-214 (Nektar).
2. Have previously undergone any of the following NMIBC-related treatments:

   1. Received extensive pelvic radiotherapy (involving >30% of bone marrow) within 2 years prior to the first dose.
   2. Received systemic therapy aimed at treating NMIBC (e.g., radiotherapy, chemotherapy, immunosuppressive therapy) within 4 weeks prior to the first dose.
   3. Received intravesical instillation aimed at treating NMIBC within 4 weeks prior to the first dose, including intravesical local treatment delivered transurethrally.
   4. Underwent TURBT or other surgical procedures targeting bladder lesions within 2 weeks prior to the first dose.

   2. Prior therapies and recovery from related toxicities：

a) Known or suspected allergy to FL115, its excipients, interleukin-based therapies, or fusion proteins (Grade 3-4), or to BCG/excipients (for Phase Ib/II).

b) Systemic immunosuppressive therapy within 4 weeks before first dose, except: ≤10 mg/day prednisone equivalent, local/inhaled/intranasal steroids, adrenal replacement ≤7.5 mg/day prednisone, or single-dose prophylaxis for contrast allergy.

c) Prior allogeneic organ or PBSC/bone marrow transplantation. d) Live virus vaccination within 4 weeks prior to first dose. e) Prior ≥ Grade 3 or treatment-discontinuation irAE due to immunotherapy, except controlled hypothyroidism, type 1 diabetes, or limited skin irAEs.

f) Unresolved AEs from prior anti-tumor therapy that have not returned to baseline or ≤ Grade 1 (per CTCAE v5.0) prior to first dose, except alopecia, ≤ Grade 2 neuropathy, or controlled hypothyroidism. Other ≤ Grade 2 AEs require PI and sponsor medical review.

3.Medical and Surgical History:

1. History or current diagnosis of muscle-invasive (T2-T4), locally advanced (T3/T4, any N), or metastatic bladder cancer.
2. History or evidence of upper urinary tract (kidney, renal pelvis, ureter) or prostatic urethral tumors.
3. Known vesicoureteral reflux or evidence of bladder perforation.
4. Active urinary tract infection.
5. Discontinuation of prior BCG therapy due to severe adverse events such as sepsis, systemic infection requiring treatment, or urinary incontinence (Phase Ib and II applicable).
6. Post-TURBT complications that preclude intravesical instillation, per investigator judgment.
7. Clinically significant polyuria (e.g., 24-hour urine volume >4000 mL).
8. History of other malignancies within 2 years prior to screening that have shown progression or required active treatment.
9. Active or prior autoimmune disease requiring systemic immunosuppressants or corticosteroids.
10. History of severe pulmonary toxicity.
11. History or imaging evidence of active pulmonary TB within 1 year prior to enrollment, or prior TB infection not adequately treated.
12. Uncontrolled pleural, pericardial, or peritoneal effusion deemed clinically significant by the investigator (e.g., requiring repeated drainage >once/month).
13. History of significant cardiovascular disease.
14. Major surgery within 4 weeks prior to signing informed consent.

    4.Infectious Disease History

a) Severe infections within 4 weeks before first dose. b) Any history of confirmed active HBV, HCV, HIV, or active tuberculosis infection.

5.Other Conditions

1. Pregnant or breastfeeding women.
2. Known, documented, or suspected substance abuse. Exceptions: Prescribed opioids for pain control or other investigator-approved, medically justified cases (pending sponsor medical lead agreement).
3. Any other conditions deemed by the investigator to render the subject unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2027-10-10 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
MTD | up to 15 months
  Maximal Tolerance Dose
RP2D | up to 15 months
  Recommended Phase II Dose
Safety and tolerability | through study completion, up to 5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Complete Response | 36 months
  Assess incidence of complete response of CIS (with or without Ta/T1 papillary disease) patients at any time
Disease-Free Rate | 12 months
  Assess disease-free rate at 12 months since first study treatment

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Fujian
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Sichuan Academy of Medical Sciences · Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Fudan University Cancer Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No
Our research is based on earlier studies and there is a high degree of uncertainty. We will consider sharing the results only after we have obtained sufficient data.